CLINICAL TRIAL: NCT04064892
Title: Physical Activity Interventions for Young Cancer Survivors
Brief Title: Physical Activity Intervention for Young Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Haus of Volta (Unknown)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 181367
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Quality of Life; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Participants will receive a 12-week, individually-tailored, video conference-based physical activity intervention
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — The intervention will use peer mentors, motivational interviewing, and technology (Fitbit, Fitbit Coach App, & Fitbit message board) to support behavior change. All participants will receive phone or video calls from their peer mentors every other week, and interact with their peer mentor and other participants through a private Fitbit message board at least weekly. Peer mentors will use Fitbit data to identify participants who need additional support to increase their activity.

SUMMARY:
The proposed mixed methods pilot study will enroll 20 young breast cancer survivors into a 12-week technology-based, remotely-delivered, peer-moderated physical activity program to examine the effects of the intervention on objectively measured physical activity and multiple aspects of quality of life; and conduct qualitative analyses to refine the intervention for a future randomized controlled trial.

DETAILED DESCRIPTION:
Young breast cancer survivors (i.e. those < 50 years old) have lower survival rates than their older counterparts and experience unique physical and mental challenges associated with their cancer treatments. Depression, anxiety, and poor body image are common in young breast cancer survivors. Research in older breast cancer survivors has shown that physical activity can decrease cancer recurrence and mortality, and improve many aspects of quality of life. Few physical activity intervention studies have been conducted in young breast cancer survivors, despite the fact that young survivors would be best served by age-specific interventions designed to target their needs. Remotely-delivered, technology-based interventions may be important to help young breast cancer survivors overcome unique barriers to increasing physical activity and improving quality of life.

The study aims are: 1) Explore the feasibility and acceptability of a technology-based, remotely-delivered, peer-moderated physical activity intervention for young breast cancer survivors; 2a) Assess the invention's impact on change in physical activity; and 2b) Measure the intervention's effect on multiple aspects of quality of life

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer between 18-49 years old
* Completed active treatment (chemotherapy, radiation) at least 6 months prior to enrollment
* Self-report low levels of moderate to vigorous physical activity each week
* Accessible by phone or video chat
* Have a Fitbit compatible cellphone, tablet, or laptop with Internet

Exclusion Criteria:

* medical condition that could make it potentially unsafe to be in an unsupervised physical activity intervention
* currently pregnant
* unable to commit to intervention schedule
* prisoner

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Baseline to 12 weeks
  The ActiGraph GT3X+ accelerometer will be used to measure change in minutes of moderate to vigorous physical activity from baseline to 12 weeks. For 7 days around each assessment time point, participants will wear the accelerometer.

SECONDARY OUTCOMES:
Body Image Scale | Baseline to 12 weeks
  The Body Image Scale will be used to measure changes in perceptions of body image from baseline to 12 weeks. Scores range from 0 to 30. A higher score indicates more distress.
Female Sexual Function Index | Baseline to 12 weeks
  The Female Sexual Function Index will be used to measure change in self-reported sexual functioning from baseline to 12 weeks. Scores range from 2 to 36. A higher score indicates fewer problems with sexual functioning.
PROMIS Cancer - Fatigue | Baseline to 12 weeks
  Change in fatigue from baseline to 12 weeks will be assessed via a Patient-Reported Outcome Measurement Information System (PROMIS) computer adaptive test (CAT), PROMIS Cancer- Fatigue. CAT items are dynamically selected for administration from an item bank based upon the respondent's previous answers. Participants will complete 4-12 items. This measure yields a T-Score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher levels of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiner LS, Nagel S, Irene Su H, Hurst S, Levy SS, Arredondo EM, Hekler E, Hartman SJ. A remotely delivered, peer-led intervention to improve physical activity and quality of life in younger breast cancer survivors. J Behav Med. 2023 Aug;46(4):578-593. doi: 10.1007/s10865-022-00381-8. Epub 2022 Dec 7. PMID 36479658
- [Derived] Weiner LS, Nagel S, Su HI, Hurst S, Hartman SJ. A Remotely Delivered, Peer-Led Physical Activity Intervention for Younger Breast Cancer Survivors (Pink Body Spirit): Protocol for a Feasibility Study and Mixed Methods Process Evaluation. JMIR Res Protoc. 2020 Jul 8;9(7):e18420. doi: 10.2196/18420. PMID 32673270